CLINICAL TRIAL: NCT07019909
Title: A Phase 1, Randomized, Double-Blind, Third-Party-Unblinded Trial to Evaluate the Safety and Immunogenicity of 20-valent Pneumococcal Conjugate Vaccine (20vPnC) and 13-valent Pneumococcal Conjugate Vaccine (13vPnC) in Pneumococcal Vaccine-Naïve Adults 50 Years of Age and Older in China
Brief Title: A Study to Learn About How Safe and Effective is 20vPnC and 13vPnC Vaccines in Chinese Adults
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: B7471039
Record Dates: First submitted 2025-06-05; First posted 2025-06-13 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Pneumococcal Disease
MeSH Terms: conditions — Pneumococcal Infections

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 20vPnC (Experimental): Single dose of 20-valent pneumococcal conjugate vaccine
  Interventions: Biological: 20vPnC
- 13vPnC (Experimental): Single dose of 13-valent pneumococcal conjugate vaccine
  Interventions: Biological: 13vPnC

INTERVENTIONS:
Biological: 20vPnC — 20 valent pneumococcal conjugate vaccine
  Arms: 20vPnC
Biological: 13vPnC — 13 valent pneumococcal conjugate vaccine
  Arms: 13vPnC

SUMMARY:
This Phase 1, randomized, double-blind, third-party-unblinded study will be conducted at investigational sites in China. The purpose of the study is to learn about the safety and immune response of 20vPnC and 13vPnC in Chinese adults 50 years of age and older who did not receive any of pneumococcal vaccine in the past

DETAILED DESCRIPTION:
The purpose of the study is to learn about the safety and immune response of 20vPnC and 13vPnC vaccines in Chinese adults. This study is seeking for participants who:

* are 50 years of age and older
* did not receive any of vaccines used to treat infections caused by the bacteria called Streptococcus pneumonia in the past.

The participants will be grouped by three age groups:

* Adults between 50 to 59 years of age
* Adults between 60 to 64 years of age
* Adults who are 65 years of age or above

All participants in this study will receive a single dose of 20vPnC or 13vPnC at study clinic. The study will look at the experiences of people receiving 20vPnC and 13vPnC. This will help decide if the study vaccine is safe.

The total duration of taking part in the study will be around 6 months, with 6 visits.

ELIGIBILITY:
Key inclusion criteria:

1.Generally healthy adults including those with preexisting stable disease determined to be eligible based on clinical assessment, medical history and clinical judgment.

Key exclusion criteria:

1. History of microbiologically-proven invasive disease caused by Streptococcus pneumoniae
2. Previous vaccination with any licensed or investigational pneumococcal vaccine or planned receipt through study participation.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2025-07-06 (Actual); Primary Completion 2026-02-03 (Estimated); Study Completion 2026-02-03 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants reporting prompted local reactions within 7 days following investigational product administration | Within 7 days after vaccination
  Prespecified local reactions (redness, swelling, and pain at the injection site)
Percentage of participants reporting prompted systemic events within 7 days following investigational product administration | Within 7 days after vaccination
  Prespecified systemic events (fever, headache, fatigue, muscle pain, and joint pain)
Percentage of participants reporting adverse events (AEs) through 1 month following investigational product administration | Within 1 month after vaccination
  Adverse events occurring within 1 month after vaccination
Percentage of participants reporting serious adverse events (SAEs) throughout the study | Within 6 months after vaccination
  SAEs occurring within 6 months after vaccination
Percentage of participants reporting abnormal hematology, biochemistry, and urinalysis and microscopy laboratory values | 3 to 5 days after vaccination
  Abnormal hematology, biochemistry, and urinalysis and microscopy laboratory values

SECONDARY OUTCOMES:
Pneumococcal serotype-specific Opsonophagocytic activity (OPA) geometric mean titer (GMT) | 1 month after vaccination
  Pneumococcal serotype-specific OPA GMTs
Pneumococcal serotype-specific OPA geometric mean fold rise (GMFR) | Before vaccination to 1 month after vaccination
  Pneumococcal serotype-specific OPA GMFRs

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (3):
- China (3):
  - Zhejiang provincial center for disease control and prevention, Hangzhou, Zhejiang
  - Kaihua County Center For Disease Prevention and Control, Kaihua, Zhejiang
  - Kaihua County Center For Disease Prevention and Control, Quzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7471039